| <b>gsk</b> GlaxoSmithKline | Stu | dy RAP |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ⊠ Final | Date: 26SEP 2008 |

# **Study Reporting and Analysis Plan**

HIV Prophylactic Vaccine

PRO HIV-005 (108706)



| GlaxoSmithKline Biologicals | | | |
|---|---|---|---|
| Global Clinical Research & Development | | | |
| Study 1 | Reporting and A | Analysis Plan Ap | proval |
| Title: | Dose-ranging stu | dy to evaluate the saf | ety and immunogenicity |
| | of GSK Biologica | als' HIV vaccine 732 | 461, adjuvanted or not, |
| | | ed as a 3 2-dose sched<br>e volunteers, aged 18 | _ |
| eTrack study number | 108706 | | |
| eTrack abbreviated | PRO HIV-005 | | |
| title | | | |
| Scope: | All Final data per | taining to the above s | study |
| Date: | 11 MAR 2008 (a | mendment 1) | |
| Co-ordinating author: | | | |
| | (Amendment 1) | | |
| | (Amendment 2) | | |
| Others author(s): | | | |
| Approved by: | | | |
| Worldwide Project | | | |
| Clinical Development<br>Manager | | | |
| _ | Name | Signature | dd-mmm-yyyy |
| Project Statistician | | | |
| - | Name | Signature | dd-mmm-yyyy |
| | PPD | | |
| Statistical Manager | Name | Signature | dd-mmm-yyyy |
| | PPD | | |



## **TABLE OF CONTENTS**

| | | | Page | |
|---|---|---|---|---|
| 1. | INTR | ODUCTIO | DN | 6 |
| 2 | CDIT | | DEVALUATION OF OR JECTIVES | 7 |
| 2. | 2.1. | | R EVALUATION OF OBJECTIVESes | |
| | 2.1. | 2.1.1. | Primary objectives | |
| | | 2.1.1. | Secondary Objectives | |
| | | 2.1.2. | Exploratory Objectives | |
| | 2.2. | | ts | |
| | 2.2. | 2.2.1. | Primary endpoints | |
| | | 2.2.2. | Secondary endpoints | |
| | | 2.2.3. | Exploratory endpoints | |
| | 2.3. | | ohorts | |
| | 2.0. | 2.3.1. | Total Vaccinated cohort | |
| | | 2.3.2. | According-To-Protocol (ATP) cohort for analysis of safety | |
| | | 2.3.3. | According-To-Protocol (ATP) cohort for analysis of | |
| | | | immunogenicity | 9 |
| | 2.4. | Group d | lescription | |
| | 2.5. | | safety analysis | |
| | | | , , | |
| 3. | STAT | ISTICAL I | METHODOLOGY AND ANALYSIS | 11 |
| | 3.1. | Study co | ohorts and demography analysis | 11 |
| | | 3.1.1. | Study cohorts | |
| | | 3.1.2. | Analysis of demographics/baseline characteristics | |
| | 3.2. | | genicity | |
| | | 3.2.1. | Cohorts | |
| | | 3.2.2. | Handling of missing data | |
| | | 3.2.3. | Compliance | |
| | | 3.2.4. | All symptoms | |
| | | 3.2.5. | Solicited symptoms | |
| | | 3.2.6. | Unsolicited symptoms | |
| | | 3.2.7. | Serious adverse events | |
| | | 3.2.8. | Haematological and biochemical parameters | |
| | | 3.2.9. | Concomitant medication | |
| | 0.0 | 3.2.10. | Exploratory analyses | |
| | 3.3. | | ogenicity | 16 |
| | | 3.3.1. | Cohorts and stratification | |
| | | 3.3.2. | Derived and transformed data | |
| | | 3.3.3. | Lab assays for immunogenicity | 18 |
| | | 3.3.4. | Handling of missing data | |
| | | 3.3.5. | Cell-mediated immune response | |
| | | | 3.3.5.1. Within group assessment | |
| | | 3.3.6. | Humoral response | |
| | | 5.5.0. | 3.3.6.1. Within group assessment | 20<br>2∩ |
| | | | o.o.o. i. within group assessine it | 20 |



|---|---|---|---|---|---|
| | 3.4. | Method | ology for co | mputing CI | 21 |
| 4. | CHAN | IGE FRO | м ркотос | OL | 22 |
| 5. | INDIV | IDUAL LI | STINGS AN | ND TABLES | 23 |
| | 5.1. | | | | |
| | 5.2. | | | | |
| | 5.3. | Templat | te of tables | | 28 |
| | | 5.3.1. | Study col | norts and demography analysis | 28 |
| | | | | Study cohorts | |
| | | | | Demographic characteristics | |
| | | 5.3.2. | | nicity/Safety | |
| | | | 5.3.2.1. | Compliance with respect to documenting safety | 32 |
| | | | 5.3.2.2. | All symptoms | |
| | | | 5.3.2.3. | Solicited symptoms | 34 |
| | | | 5.3.2.4. | Unsolicited symptoms | 37 |
| | | | 5.3.2.5. | Serious adverse events | |
| | | | 5.3.2.6. | Haematology and biochemistry | 39 |
| | | | 5.3.2.7. | Concomitant medications | 40 |
| | | 5.3.3. | Immunog | enicity | 41 |
| | | | 5.3.3.1. | CD4+/CD8+ T-cells response by ICS | 41 |
| | | | 5.3.3.2. | Antibodies | 43 |

# Study RAP Study Id: 108706 Abbreviated Title: PRO HIV-005 Version: Draft version Image: Property of the property of the prop

# CONFIDENTIAL LIST OF ABBREVIATIONS

**AE** Adverse event

**ATP** According to Protocol

**BCSP** Biologicals clinical safety and pharmacovigilance

**CD40L** Immune cells that carry a marker on its surface known as Cluster of

Differentiation 40L Immune cells that carry a marker on its surface

known as Cluster of Differentiation 40L

CI Confidence Interval

**CMI** Cell-mediated immunity

**ELISA** Enzyme Linked Immunosorbent Assay

GCRD Global clinical research and developpement

**GMT** Geometric mean titer

**GSK** GlaxoSmithKline

**MedDRA** Medical Dictionary for Regulatory Activities

RAP Report analysis plan

**SAE** Serious adverse event

**SRT** Safety review team

| <b>gsk</b> GlaxoSmithKline | Stu | dy RAP |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

# 1. INTRODUCTION

The purpose of this document is to describe (on the basis of protocol/amendment dated 08 October 2007):

- criteria for evaluation of objectives in terms of endpoints, study cohorts, derived data, group description and interim analysis (paragraph 2);
- statistical methodology and planned analyses (paragraph 3);
- change(s) from protocol (paragraph 4);
- individual listings, list of tables and template tables (paragraph 5).

Any planned modification of the statistical analyses should be documented by an amendment to the RAP (Table 1).

Table 1. List of amendments to the RAP

| Date | Description |
|---|---|
| 28 JAN 2008 | First version |
| 18 FEB 2008 | Amendment 1 |
| | cut-off definition for CD4/CD8 |
| | modification of CD8 exploratory endpoints |
| | Correction of grading for exploratory safety analysis |
| | N definition for CMI responders |
| 26SEP2008 | Amendement 2 |
| | Precisions for final analysis (month 12 data available): |
| | ATP cohort definition clarified |
| | Group order has been modified to account for the order actually used in the presentations |

| gsk GlaxoSmithKline | St | udy RAP |
|-------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft versio | n ⊠ Final | Date: 26SEP 2008 |

#### 2. CRITERIA FOR EVALUATION OF OBJECTIVES

# 2.1. Objectives

# 2.1.1. Primary objectives

- To evaluate the reactogenicity and safety of the candidate vaccine F4co (p24-RT-Nef-p17) with or without AS01B adjuvant at three different doses (10-30-90 μg).
- To evaluate the CD4+ T-cell response to the candidate vaccine F4co (p24-RT-Nefp17) with or without AS01B at three different doses (10-30-90 μg) in terms of proportion of responders to at least 1, 2, 3 antigens and to all 4 antigens determined two weeks after the second vaccination

# 2.1.2. Secondary Objectives

- To evaluate the CD4+ T-cell immune response to the candidate vaccine F4co (p24-RT-Nef-p17) with or without AS01B at three different doses (10-30-90 μg) after two vaccinations.
- To evaluate the serological response to the candidate vaccine F4co (p24-RT-Nefp17) with or without AS01B at three different doses (10-30-90 μg) after two vaccinations
- To evaluate the persistence of cell-mediated and serological responses to the candidate vaccine F4co (p24-RT-Nef-p17) with or without AS01B at three different doses (10-30-90 µg).

# 2.1.3. Exploratory Objectives

- To evaluate the cross clades reactivity determined by ICS 2 weeks and/or 1 month after the second vaccination.
- To evaluate the CD8+ T-cells immune response to the candidate vaccine F4co (p24-RT-Nef-p17) with or without AS01B at three different doses (10-30-90 μg).

# 2.2. Endpoints

# 2.2.1. Primary endpoints

#### Reactogenicity and safety

- Occurrence, intensity and relationship to vaccination of solicited local and general symptoms during a 7-day (Day 0 to Day 6) follow-up period after each vaccination.
- Occurrence, intensity and relationship to vaccination of unsolicited symptoms during a 30-day (Day 0 to Day 29) follow-up period after each vaccination.

| <b>gsk</b> GlaxoSmithKline | Stu | dy RAP |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | n ⊠ Final | Date: 26SEP 2008 |

- Occurrence and relationship to vaccination of serious adverse events during the whole study period.
- Haematological and biochemical levels at months 0, 1, 2, 6, 9, 12 and at Day 44 (two weeks after the second vaccination) in all subjects.

#### **Immunogenicity**

 Frequency of CD4+ T cells expressing at least two cytokines including IL-2 equal or above the cut-off to at least 1, 2, 3 antigens and to all 4 antigens at Day 44 (two weeks after the second vaccination).

# 2.2.2. Secondary endpoints

- Frequency of p17, p24, Nef and RT-specific CD4+ T cells expressing IL-2 and/or TNF-α and/or IFN-γ and/or CD40-L, as determined by ICS at Months 0, 2, 6, 12 and at Day 44 (two weeks after the second vaccination).
- Frequency of p17, p24, Nef and RT-specific CD4+ T cells expressing at least 2 cytokines including IL-2 equal or above the cut-off at Months 0, 2, 6, 12 and at Day 44 (two weeks after the second vaccination).
- Antibody titers to p17, p24, Nef, RT and F4co as measured by ELISA at Months 0,
   2, 6, 12 and at Day 44 (two weeks after the second vaccination).

# 2.2.3. Exploratory endpoints

- Frequency of p17, p24, Nef and RT-specific CD4+ T cells to other HIV clades expressing IL-2 and/or TNF-α and/or IFN-γ and/or CD40-L, as determined by ICS at Day 44 (two weeks after the second vaccination) and/or at Month 2.
- Frequency of p17, p24, Nef and RT-specific CD8+ T cells expressing HL-2 and/or TNF-α and/or IFN-γ and/or CD40 L, as determined by ICS at Months 0, 2, 6, 12 and at Day 44 (two weeks after the second vaccination) (amendment 1).
- Frequency of p17, p24, Nef and RT-specific CD8+ T cells expressing at least 2 cytokines (H-2 and/or TNF-α and/or IFN-γ and/or CD40-L) equal or above the cutoff at Months 0, 2, 6, 12 and at Day 44 (two weeks after the second vaccination) (amendment 1).

# 2.3. Study cohorts

Three cohorts will be evaluated, as described below.

#### 2.3.1. Total Vaccinated cohort

The Total Vaccinated cohort will include all vaccinated subjects.

| gsk GlaxoSmithKline | Stu | dy RAP |
|--------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

Thus, the Total Vaccinated cohort for analysis of safety will include all subjects with at least one vaccine administration documented. This is valid for both Month 2 and Month12 analyses

The Total Vaccinated cohort for analysis of immunogenicity will include vaccinated subjects for whom data concerning immunogenicity endpoint measures are available. This is valid for both Month 2 and Month 12 analyses

The Total Vaccinated cohort analysis will be performed per treatment actually administered. This is valid for both Month 2 and Month 12 analyses

# 2.3.2. According-To-Protocol (ATP) cohort for analysis of safety

The ATP cohort will include all vaccinated subjects

- who have received at least one dose of study vaccine according to their random assignment.
- with sufficient data to perform an analysis of safety (at least one dose with safety follow-up).
- for whom administration route of study vaccines is known.
- who have not received a vaccine not specified or forbidden in the protocol. This
  criterion would potentially lead to a different ATP cohort for Month 2 and for Month
  12 analyses.
- for whom the randomization code has not been broken. This criterion would potentially lead to a different ATP cohort for Month 2 and for Month 12 analyses.

It has been decided to present the results for Month 6 and Month 12 based on the Month 12 cohort definition, while all results produced at Month 2 analysis will be based on Month 2 cohort.

# 2.3.3. According-To-Protocol (ATP) cohort for analysis of immunogenicity

The ATP cohort for analysis of immunogenicity will include all evaluable subjects, (i.e., those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity endpoint measures are available. This definition would potentially lead to a different ATP cohort for Month 2 and for Month 12 analyses.

It has been decided to present the results for Month 6 and Month 12 based on the Month 12 cohort definition, while all results produced at Month 2 analysis will be based on Month 2 cohort

| gsk | | Study RAP |
|----------------------|-------------------|------------------|
| Study ld: 108706 | Abbreviated Title | tle: PRO HIV-005 |
| Version: Draft versi | on ⊠ Final | Date: 26SEP 2008 |


# 2.4. Group description

The following group description will be used for the demography, reactogenicity and immunogenicity analyses.

| Group order in tables | Group label in tables (8 characters only) | Group definition for footnote |
|---|---|---|
| 1 | F4co10W | F4co 10 µg + WFI |
| 2 | F4co30W | F4co 30 µg + WFI |
| 3 | F4co90W | F4co 90 µg + WFI |
| 4 | F4co10A | F4co 10 µg + AS01B |
| 5 | F4co30A | F4co 30 µg + AS01B |
| 6 | F4co90A | F4co 90 µg + AS01B |

| gsk GlaxoSmithKline | Stu | idy RAP |
|------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

# 2.5. Interim safety analysis

Six interim analyses were planned for safety evaluation (see Section 5.6).

These analyses have been performed at the end of the 7-day follow-up period (Days 7 and 37) after each vaccine injection in a subset of 12 subjects and for each vaccine dose (10, 30 and 90  $\mu$ g).

Analysis has been done on uncleaned and blinded data. Individual data listings of the demographic and safety data (solicited/unsolicited AE, SAE, haematology and biochemistry values) have been provided to the SRT. Tables with the number of subjects responding to each stopping rules have been also provided.

No clinical report has been written.

As interim safety analyses have been already performed, description of tables and template will be not be part of a RAP.

Protocol forwarded that Final analysis would be performed in 2 steps:

- A first analysis was performed on all data up to and including month 2. These analyses were based on amendment 2 of the present document.
- A second analysis was planned for the report to be written at the end of the study (month 12). The analyses to be covered are detailed in this version of the RAP.

#### 3. STATISTICAL METHODOLOGY AND ANALYSIS

# 3.1. Study cohorts and demography analysis

# 3.1.1. Study cohorts

The number and percentage of subjects included in each of the study cohorts, for both the Month 2 and thre Month 12 analyses, as well as the reason(s) for elimination will be presented.

The number of subjects who attended each study visit and the identification numbers of subjects who dropped out from the study along with the reason for withdrawal will be displayed per group for both study conclusions (month 2 and month 12). From an analysis perspective, a "drop-out" is any subject who did not come back for the concluding visit/contact foreseen in the protocol. A subject who returns for the concluding visit/contact foreseen in the protocol is considered to have completed the study. Reasons for drop-out from the study will also be summarised by group.

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | n ⊠ Final | Date: 26SEP 2008 |

The age at the first vaccination and the intervals between visits defined in the protocol should be followed as closely as possible. Subjects falling outside of these intervals will be reviewed and eventually excluded from the According-To-Protocol immunogenicity analysis:

| Interval | Length of interval (Days) |
|-------------------|---------------------------|
| Visit 2 → Visit 3 | 14 ± 2 |
| Visit 2 → Visit 4 | 30 - 34 |
| Visit 1 → Visit 5 | $180 \pm 14$ |
| Visit 5 → Visit 7 | $180 \pm 14$ |

The number and percentage of subjects out of these defined limits for the age and/or the intervals between visits will be described. The denominator used to calculate the percentage is the number of subjects present at the considered visits.

An overview of the number of vaccine doses received will be displayed (only for Month 2 analysis).

For each activity, the minimum and maximum dates over all vaccinated subjects will be presented.

# 3.1.2. Analysis of demographics/baseline characteristics

Demographic characteristics (age, gender, race) of each study cohort, for both the Month 2 and thre Month 12 analyses, will be tabulated.

The mean age (plus range and standard deviation) by gender of the enrolled subjects, as a whole, and per group, will be calculated, (only for Month 2 analysis).

# 3.2. Reactogenicity

#### 3.2.1. Cohorts

The primary analysis will be based on the total vaccinated cohort. If the percent of enrolled subjects excluded from the ATP cohort for analysis of safety is more than 5%, a second analysis based on this ATP cohort will be performed to complement the Total analysis.

#### 3.2.2. Handling of missing data

For the analysis of solicited symptoms, missing or non-evaluable measurements will not be replaced. Therefore the analysis of the solicited symptoms based on the

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | n ⊠ Final | Date: 26SEP 2008 |

totalvaccinated cohort will include only subjects/doses with documented safety data (i.e.symptom screen/sheet completed).

For the analysis of unsolicited adverse events/serious adverse event/concomitant medication, all vaccinated subjects will be considered and subjects who did not report an event will be considered as subjects without an event.

# 3.2.3. Compliance

This analysis will be performed for Month 2 only.

The number of doses injected, the number of doses not given according-to-protocol, the number of symptom sheets (SS) transcribed for local and general symptoms and, the compliance for local and general symptoms will be tabulated. Compliance (%) is defined as the number of (local/general) symptom sheets completed divided by the number of doses administered for a specified group. The number of doses not given according-to-protocol is the number of doses administered at wrong site and/or side, or administered using a wrong route as compared to the protocol specifications.

## 3.2.4. All symptoms

This analysis will be performed for Month 2 only.

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the solicited follow-up period (Day 0 to Day 6) will be tabulated with exact 95% confidence interval (CI) after each vaccine injection and overall.

The percentage of vaccine injections followed by at least one local AE (solicited and unsolicited), by at least one general AE (solicited and unsolicited) and by any AE will be tabulated, overall vaccination course, with exact 95% CI.

# 3.2.5. Solicited symptoms

This analysis will be performed for Month 2 only.

The number and percentage of subjects reporting each individual solicited local and general AE during the solicited follow-up period will be tabulated with exact 95% CI.

The number and percentage of vaccine injections followed by each individual solicited local and general AE will be tabulated, overall vaccination course, with exact 95% CI.

| gsk | SmithKline | Study RAP | |
|-----------|-----------------|--------------------|------------------|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | | Date: 26SEP 2008 |

The maximum intensity of fever and local injection site redness/swelling will be scored as follows:

| Symptoms | Grade | Scale |
|--------------------------------|-------|------------------|
| Fever | 0 | ] 37.5°C |
| (Oral or Axillary temperature) | 1 | [37.5°C – 38°C] |
| , | 2 | ] 38°C - 39°C ] |
| | 3 | [39°C |
| Redness/Swelling | 0 | 0 mmm |
| | 1 | [ 20 mm |
| | 2 | ]20 mm – 50 mm ] |
| | 3 | ] 50 mm |

The same tabulations will be done for grade 3 adverse events and/or for adverse events with relationship to vaccination.

The number and percentage of of subjects reporting a solicited symptom will be also presented by duration ( $\leq 2$  days or > 2 days).

For fever, temperatures will be also summarized in 0.5°C increments.

The number of days with a solicited symptom during the solicited follow-up period will be aslo presented. The same tabulations will be done for grade 3 adverse events and/or for adverse events with relationship to vaccination.

## 3.2.6. Unsolicited symptoms

This analysis will be performed for Month 2 only.

The proportion of subjects with at least one report of unsolicited AE classified by the Medical Dictionary for Regulatory Activities (MedDRA) and reported up to 30 days after vaccination will be tabulated with exact 95% CI.

The same tabulations will be done for grade 3 adverse events and/or for adverse events with relationship to vaccination.

#### 3.2.7. Serious adverse events

Serious AEs and withdrawal due to AEs will be described in detail for both the Month 2 and thre Month 12 analyses.

| gsk GlaxoSmithKline | Study RAP | |
|--------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

# 3.2.8. Haematological and biochemical parameters

The frequency distribution of values below, within and above normal ranges will be tabulated per treatment group at each scheduled time point. In addition, change from baseline will be also tabulated.

Cleaning for these data for the month 12 analysis will only performed in a second step. This has no impact on the other analyses to be performed, as these data will not impact on the cohort definition.

#### 3.2.9. Concomitant medication

This analysis will be performed for Month 2 only.

The number and percentage of subjects with concomitant medication(s), with antipyretics, with antibiotics and with immunosuppressant within 30 days post-vaccination will be tabulated with exact 95% CI. Concomitant medications will be classified in antipyretics, antibiotics and immunosuppressant according to the WHO drug dictionary.

# 3.2.10. Exploratory analyses

Analyses of solicited symptoms will be also performed with the following grading to facilitate comparisons with other GSK studies:

| Symptoms | Grade | Scale |
|--------------------------------|-------|-------------------|
| Fever | 0 | ] 38°C |
| (Oral or Axillary temperature) | 1 | [ 38°C – 38.5°C [ |
| | 2 | [ 38.5°C – 39°C [ |
| | 3 | [39°C – 40°C [ |
| | 4 | [40°C |
| Redness/Swelling | 0 | ≤ 20 <b>0</b> mm |
| | | (amendment 1) |
| | 1 | ]20 mm – 50 mm] |
| | 2 | ]50 mm – 100 mm ] |
| | 3 | ] 100 mm |

| gsk | SmithKline | Study RAP | |
|-----------|-----------------|--------------------|------------------|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | ☑ Final | Date: 26SEP 2008 |

# 3.3. Immunogenicity

#### 3.3.1. Cohorts and stratification

The primary analysis will be based on the ATP cohort for analysis of immunogenicity. If the percent of enrolled subjects excluded from this ATP cohort is more than 5%, a second analysis based on the Total Vaccinated cohort will be performed to complement the ATP analysis.

It has been decided to present the results for Month 6 and Month 12 based on the Month 12 cohort definition, while all results produced at Month 2 analysis will be based on Month 2 cohort. For clarity purposes, Month 12 analyses which include only descriptive summaries will be presented in separate tables with only the relevant time points included (Month 6 and Month 12).

#### 3.3.2. Derived and transformed data

## Serology data

- The cut-off values for antibody titers will be defined by the laboratory before the analysis.
- A seronegative subject is a subject whose titer is below the cut-off value.
- A seropositive subject is a subject whose titer is greater than or equal to the cut-off value.
- The seropositivity rate is defined as the percentage of seropositive subjects.
- The Geometric Mean Titers (GMTs) calculations will be performed by taking the
  anti-log of the mean of the log titer transformations. Antibody titers below the cut-off
  of the assay will be given an arbitrary value of half the cut-off for the purpose of
  GMT calculation.

#### ICS data

- ICS data will be expressed as antigen-specific CD4+/CD8+ T-cells per million respectively of CD4+ or CD8+ T-cells.
- The cut-off will be choosen on the basis of pre-vaccination response for all subjects, by examining percentiles (95th percentile included) of the different antigens and the different cytokines (amendment 1). A 95<sup>th</sup> percentile will be determined for each antigen on the CD4 expressing at least two cytokines (all doubles) for CD4 responses and on the CD8 expressing at least one cytokine for CD8 responses.

| gsk | Study RAP | |
|----------------------|-------------------|------------------|
| Study ld: 108706 | Abbreviated Title | tle: PRO HIV-005 |
| Version: Draft versi | on ⊠ Final | Date: 26SEP 2008 |

The cut-off will be defined as the rounded (superior hundred) maximum 95th percentile among the 4 antigens (amendment 1).

- A responder is a subject with antigen-specific CD4+/CD8+ T-cells response greater than or equal to the cut-off value.
- Frequency of CD4+/CD8+ T-cells expressing cytokines to the fusion protein F4co (all antigens) will be estimated by adding individual frequencies of CD4+/CD8+ T-cells to each 4 antigens (p17, p24, Nef, RT).

| gsk GlaxoSmithKline | Study RAP | |
|------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

## 3.3.3. Lab assays for immunogenicity

The following table describes the lab assays that will be analyzed for immune response:

| Assay | Assay<br>method | Test kit/<br>Manufacturer | Assay unit | Assay<br>cut-off or<br>Limit of<br>detection | Laboratory |
|---|---|---|---|---|---|
| Anti-p17,-24,-RT,-<br>Nef, -F4co antibodies | ELISA | In-house ELISA | EU/mL | To be determined | CEVAC,<br>Belgium |
| p17-,24-,RT-,Nef-<br>specific effector<br>T-cells | Flow<br>Cytometry,<br>ICS | In-house ICS | Number of<br>cytokine(s)<br>positive cells<br>per 10 <sup>6</sup> cells | To be determined | *CEVAC,<br>Belgium |

<sup>\*</sup> Or GSK Biologicals,

# 3.3.4. Handling of missing data

For a given subject and a given immunogenicity measurement, missing or non-evaluable measurements will not be replaced.

For the calculation of percentage of responders to 1, 2, 3 and all 4 antigens, subjects with missing data to at least one of the concerned antigen(s) will not be taken into account.

## 3.3.5. Cell-mediated immune response

#### 3.3.5.1. Within group assessment

#### CD4+ and CD8+ T-cells response

For cell-mediated immune response, the following parameters will be tabulated by vaccine groups at months 0, 2, 6, 12 and at day 44 (two weeks after the second vaccination):

- descriptive statistics of the frequency of CD4+/CD8+ T cell expressing at least two different cytokines (IFN-γ, IL-2, TNF-α,CD40L) to each antigen and to all antigens;
- descriptive statistics of the frequency of CD4+/CD8+ T cell expressing at least IFN-γ and another cytokine (IL-2, TNF-α,CD40L) to each antigen and to all antigens;
- descriptive statistics of the frequency of CD4+/CD8+-T cell expressing at least IL-2 and another cytokine (IFN-γ, TNF-α,CD40L) to each antigen and to all antigens;
- descriptive statistics of the frequency of CD4+/CD8+ T cell expressing at least TNFα and another cytokine (IFN-γ, IL-2,CD40L) to each antigen and to all antigens;
- descriptive statistics of the frequency of CD4+ T cell expressing at least CD40L and another cytokine (IFN-γ, IL-2, TNF-α) to each antigen and to all antigens.

| gsk | SmithKline | Study RAP | |
|-----------|-----------------|--------------------|------------------|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | ☑ Final | Date: 26SEP 2008 |

#### CD4+ T-cells expressing IL-2 and another cytokine

For CD4+ T-cells expressing IL-2 and another cytokine response, the following parameters will be tabulated by vaccine groups at months 0, 2, 6, 12 and at day 44 (two weeks after the second vaccination):

- percentage of responders to each antigen (p17, p24, Nef, RT);
- percentage of responders to at least one antigen (p17, p24, Nef or RT);
- percentage of responders to at least two antigens;
- percentage of responders to at least three antigens;
- percentage of responders to all four antigens (p17, p24, Nef and RT).

In addition, percentage of responders to one, two, three and four antigens will be tabulated, with and without specification of antigens.

CD8+ T-cells expressing at least 2 cytokines (HL-2 and/or TNF- $\alpha$  and/or IFN- $\gamma$  and/or CD40-L) (amendment 1)

For CD8+ T-cells, the following parameters will be tabulated by vaccine groups at months 0, 2, 6, 12 and at day 44 (two weeks after the second vaccination):

- descriptive statistics of the frequency of CD8+ T cell expressing at least one cytokine (IFN-γ and/or TNF-α) to each antigen and to all antigens
- descriptive statistics of the frequency of CD8+ T cell expressing only TNF- $\alpha$  to each antigen and to all antigens
- descriptive statistics of the frequency of CD8+ T cell expressing only IFN-γ to each antigen and to all antigens
- descriptive statistics of the frequency of CD8+ T cell expressing IFN-γ and TNF-α to each antigen and to all antigens
- for CD8+ T-cells expressing at least one cytokine, percentage of responders to each antigen (p17, p24, Nef, RT) (amendment 1)

#### 3.3.5.2. Between group assessment

For the following analyses, statistically significant differences (p-value  $\leq$  0.05) should be interpreted with caution as adjustment for multiplicity of endpoints and clinical relevance of the difference will not considered.

| gsk GlaxoSmithKline | Study RAP | |
|--------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

#### Analysis of frequency of CD4+ T-cells

A two-way ANOVA test will be performed on frequency of CD4+ T-cells expressing at least IL-2 to compare three doses of antigen F4Co with or without adjuvant two weeks after the second vaccination. The ANOVA model will include the doses (10  $\mu$ g, 30  $\mu$ g and 90  $\mu$ g) and the "adjuvants" (AS01B and WFI) as fixed effects.

If requires, the analysis will be performed on log10 frequency of CD4+ T-cells.

If interaction between doses and "adjuvant" is significant (p-value  $\leq 0.05$ ), comparison of doses will be done by "adjuvant" factor.

If difference between the three doses is significant (p-value  $\leq$  0.05), multiple comparisons will be performed and relationship between doses and CD4+ T-cell response will be also assessed.

ANOVA analyses will be done for each antigen (p17, p24, RT, Nef) and for the fusion protein F4Co.

#### Analysis of responders in terms of CD4+ T-cells

A logistic regression will be performed on occurrence of responders in terms of CD4+ T-cells expressing at least IL-2 (dichotomous response, 0 or 1) to compare three doses of antigen F4Co with or without adjuvant two weeks after the second vaccination. Doses, "adjuvant" and interaction will be included in the logistic model.

If interaction between doses and "adjuvant" is significant (p-value  $\leq$  0.05), a logistic regression will be applied by "adjuvant" factor.

Logisitic regressions will be done for responders to at least one, two, three and 4 antigens (p17, p24, RT or/and Nef).

# 3.3.6. Humoral response

#### 3.3.6.1. Within group assessment

For humoral immune response, the following parameters will be tabulated by vaccine groups for each antigen (p17, p24, Nef, RT and F4co) at months 0, 2, 6, 7, 12 and at day 44 (two weeks after the second vaccination):

- Geometric mean titers (GMTs) with 95% confidence intervals (CIs);
- Seropositivity rates with exact 95% CIs.

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | n ⊠ Final | Date: 26SEP 2008 |

# 3.4. Methodology for computing CI

All CI will be 2 sided 95% CI.

- The exact 95% CIs for a proportion within a group will be calculated from Proc StatXact [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].
- The 95% CI for geometric mean titers/concentrations (GMTs/GMCs) will be obtained within each group separately. The 95% CI for the mean of log-transformed titer/concentration will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The 95% CI for the GMTs/GMCs will be then obtained by exponential-transformation of the 95% CI for the mean of log-transformed titer/concentration.

21

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

#### 4. CHANGE FROM PROTOCOL

The cut-off will be choosen on the basis of pre-vaccination response for all subjects, by examining percentiles (95<sup>th</sup> percentile included) of the different antigens and the-different cytokines (amendment 1). A 95<sup>th</sup> percentile will be determined for each antigen on the CD4 expressing at least two cytokines (all doubles) for CD4 responses and on the CD8 expressing at least one cytokine for CD8 responses. The cut-off will be defined as the rounded (superior hundred) maximum 95th percentile among the 4 antigens (amendment 1).

To avoid a bias of analyses, cut-off will be determined for each antigens and each cytokines before the start of immunogenicity analyses (i.e, at the time of the pre-analysis meeting) on the basis of pre-vaccination blinded data (amendement 1).

In addition to analyses described in the protocol for CD4+ T-cells expressing IL-2 and another cytokine:

- percentage of responders to one, two, three and four antigens will be tabulated, with and without specification of antigens;
- a between assessment group will be performed (see section 3.3.5.2)

Cytokines measured for CD8+ T-cells response have been reduced to TNF- $\alpha$  and/or IFN- $\gamma$  (amendment 1).

The stepwise nature of the final analysis implied the use of a different cohort (called month 12 cohort) for the time points Month 6 and month 12 to account for the elimination of subjects between month 2 and month 12. It was agreed to use this Month 12 cohort for the SAE description and for the descriptive immunogenciity analysis. For this last type of analysis (immunogenciity), to avoid any possible confusion, tables for these month 6 and month 12 time points will be separate as those presented for the month 2 analysis for all preceding tilme points.

| gsk GlaxoSmithKline | Study RAP | |
|------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

# 5. INDIVIDUAL LISTINGS AND TABLES

# 5.1. Individual listings

Appendix Table I.A - Elimination codes

Appendix Table I.B - Demography

Appendix Table I.Ci - Dates of birth, Informed consent, Vaccination and blood sampling, Contact

Appendix Table I.Cii - Reason for visit not done

Appendix Table I.D - General medical history

Appendix Table I.E - Study conclusion

Appendix Table I.I - Reason for non administration of vaccine

Appendix Table II.A - Solicited local symptoms

Appendix Table II.B - Solicited general symptoms

Appendix Table II.Ci - Unsolicited adverse events within 31 days post-vaccination

Appendix Table II.Cii - Unsolicited adverse events after 31 days post-vaccination

Appendix Table II.Di - Concomitant medication

Appendix Table II.Dii - Concomitant vaccination

Appendix Table III.A - Immunogenicity (antibody response)

Appendix Table III.B - Immunogenicity (Cell-mediated immune response)

Appendix Table IV.A - Haematology

Appendix Table IV.B - Biochemistry

23

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | n ⊠ Final | Date: 26SEP 2008 |

# 5.2. List of tables

The following table summarizes all tables that will be produced for the planned interim (x for first interim analysis, xx for second interim analysis) and final analyses (see previous sections for detazils of cohort/analysis and time points):

| Denomination | Template table | Total<br>vaccinated<br>cohort | ATP cohort for immunogenicity | Macro |
|---|---|---|---|---|
| Parameter setting in stat batches | | Elim = 9 | Elim = 2 | |
| 1. Study cohorts and demography analysis | | | | |
| 1.1. Study cohorts | | | | |
| Table D - 1 Number of subjects enrolled into the study as well as the number excluded from ATP analyses with reasons for exclusion. | Template Table<br>D - 1 | Table D.0-1<br>( <i>Elim</i> = 0) | | %ELIMLIST |
| Table D - 2 Number of subjects at each visit and list of withdrawn subjects | Template Table<br>D - 2 | Supplementary<br>Table D.9-2 | | %DROPOUT |
| Table D - 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal | Template Table<br>D - 3 | Table D.9-3 | | %DROP_SUM |
| Table D - 4 Minimum and maximum activity dates | Template Table<br>D - 4 | Working Table<br>D.9-4 | | %DATE |
| Table D - 5 Number and percentage of subjects who received vaccine dose(s) | Template Table<br>D - 5 | Table D.9-5 | | %EXPO |
| Table D - 6 Deviations from specifications for age and intervals between study visits | Template Table<br>D - 6 | Supplementary<br>Table D.9-6 | | %INT_VAL |
| 1.2. Demographic characteristics | | | | |
| Table D – 7 Summary of demographic characteristics | Template Table<br>D - 7 | Table D.9-7 | Table D.9-8b | %DEMOGRA |

24



|---|---|---|---|---|
| Denomination | Template table | Total<br>vaccinated<br>cohort | ATP cohort for immunogenicity | Macro |
| 2. Reactogenicity/safety analysis | | | | |
| 2.1. Compliance | | | | |
| Table R - 1 Compliance in returning symptom | Template Table | Working Table | | %COMPLI |
| sheets | R-1 | R.9-1 | | 70COIVIFLI |
| Table R - 2 Compliance to data capture | Template Table<br>R - 2 | Table R.9-2 | | %CAPTURE |
| 2.2. All symptoms | | | | |
| Table R – 3.1 Incidence and nature of symptoms (solicited and unsolicited) reported during the 7 days (Days 0-6) follow-up period after each dose and overall | Template Table<br>R - 3 | Table R.9-3.1 | | %LOCGEN |
| Table R – 3.2 Incidence and nature of <b>grade 3</b> symptoms (solicited and unsolicited) reported during the 7 days (Days 0-6) follow-up period after each dose and overall | Template Table<br>R - 3 | Table R.9-3.2 | | %LOCGEN |
| Table R – 3.3 Incidence and nature of symptoms (solicited and unsolicited) with causal relationship to vaccination, reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall | Template Table<br>R - 3 | Supplementary<br>Table R.9-3.3 | | %LOCGEN |
| Table R – 3.4 Incidence and nature of <b>grade 3</b> symptoms (solicited and unsolicited) <b>with causal relationship</b> to vaccination, reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall | Template Table<br>R - 3 | Supplementary<br>Table R.9-3.4 | | %LOCGEN |
| 2.3. Solicited symptoms | | | | |
| Table R – 4 Incidence of solicited <b>local</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall | Template Table<br>R - 4 | Table R.9-4 | | %FREQ |
| Table R – 5 Incidence of solicited <b>general</b> symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall | Template Table<br>R - 5 | Table R.9-5 | | %FREQ |
| Table R – 6.1 Number of days with symptoms during the solicited post-vaccination period | Template Table<br>R - 6 | Table R.9-6.1 | | %SYMPDUR |
| Table R – 6.2 Number of days with <b>grade 3</b> symptoms during the solicited post-vaccination period | Template Table<br>R - 6 | Table R.9-6.2 | | %SYMPDUR |
| Table R – 6.3 Number of days with <b>related</b> symptoms during the solicited post-vaccination period | Template Table<br>R - 6 | Supplementary<br>Table R.9-6.3 | | %SYMPDUR |
| Table R – 6.4 Number of days with <b>Related</b> grade 3 symptoms during the solicited post-vaccination period | Template Table<br>R - 6 | Supplementary<br>Table R.9-6.4 | | %SYMPDUR |
| Table R – 7 Maximum temperature per dose, overall doses, overall subject (0.5° increments) | Template Table<br>R - 7 | Table R.9-7 | | %FREQ |



# **Study RAP**

Study Id: 108706 Abbreviated Title: PRO HIV-005

 Version:
 ☐ Draft version
 ☒ Final
 Date:
 26SEP 2008

# CONFIDENTIAL

| Denomination | Template table | Total<br>vaccinated<br>cohort | ATP cohort for immunogenicity | Macro |
|---|---|---|---|---|
| 2.4. Unsolicited symptoms | | | | |
| Table R – 8.1 Percentage of <b>subjects</b> reporting the occurrence of unsolicited symptoms classified by MEDDRA Primary System Organ Class and Preferred Term, within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 8 | Table R.9-8.1 | | %UNSOL |
| Table R – 8.2 Percentage of <b>doses</b> with unsolicited symptoms classified by MEDDRA Primary System Organ Class and Preferred Term, within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 9 | Table R.9-8.2 | | %UNSOL |
| Table R – 8.3 <b>Global Summary</b> of unsolicited signs and symptoms reported within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 10 | Table R.9-8.3 | | %UNSOL |
| Table R – 9.1 Percentage of <b>subjects</b> reporting the occurrence of <b>grade 3</b> unsolicited symptoms classified by MEDDRA Primary System Organ Class and Preferred Term, within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 8 | Table R.9-9.1 | | %UNSOL |
| Table R – 9.2 Percentage of <b>doses</b> with <b>grade</b> 3 unsolicited symptoms classified by MEDDRA Primary System Organ Class and Preferred Term, within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 9 | Table R.9-9.2 | | %UNSOL |
| Table R – 9.3 <b>Global Summary</b> of <b>grade 3</b> unsolicited signs and symptoms reported within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 10 | Table R.9-9.3 | | %UNSOL |
| Table R – 10.1 Percentage of <b>subjects</b> reporting the occurrence of unsolicited symptoms classified by MEDDRA Primary System Organ Class and Preferred Term <b>with causal relationship</b> to vaccination, within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 8 | Supplementary<br>Table R.9-10.1 | | %UNSOL |
| Table R – 10.2 Percentage of <b>doses</b> with unsolicited symptoms classified by MEDDRA Primary System Organ Class and Preferred Term <b>with causal relationship</b> to vaccination, within the 30-day (Days 0-29) post-vaccination period | Template Table<br>R - 9 | Supplementary<br>Table R.9-10.2 | | %UNSOL |
| Table R – 10.3 Global Summary of unsolicited signs and symptoms reported with causal relationship to vaccination, within the 30-day (Days 0-29) post-vaccination period 2.5. Serious adverse events | Template Table<br>R - 10 | Supplementary<br>Table R.9-10.3 | | %UNSOL |
| Table R – 11 Listing of SAEs reported during the whole study period 2.6. Haematology and biochemistry | Template Table<br>R - 11 | Table R.9-11 | | %SAE |
| Table R – 12.1 Distribution of haematology and biochemistry with respect to normal laboratory ranges | Template Table<br>R - 12 | Supplementary<br>Table R.9-12.1 | | %LAB_RW |



| Version: ☐ Draft version 区 | l Final | Date: | 26SEP 2008 | |
|---|---|---|---|---|
| Denomination | Template table | Total<br>vaccinated<br>cohort | ATP cohort for immunogenicity | Macro |
| Table R – 12.2 Change from baseline in haematological and biochemical levels with respect to normal ranges | Template Table<br>R - 1 | Supplementary<br>Table R.9-12.2 | | |
| 2.7. Concomitant medication Table R – 13 Incidence of concomitant medication during the 30-day (Days 0-29) post-vaccination period by dose and overall | Template Table<br>R - 14 | Supplementary<br>Table R.9-13 | | %CMED_INC |
| 3. Immunogenicity tables | | | | |
| 3.1. CD4+/CD8+ T-cells response by ICS Table I – 1a Frequency of CD4+ T-cells expressing cytokines (by ICS) at pre- vaccination: percentiles (amendment 1) | Template Table<br>I - 1 | | Working Table<br>I.2-1a | Specific |
| 3.1.1. Primary objective Table I – 2 CD4+ T cells expressing at least 2 cytokines including IL-2: Number and percentage of responders to at least one, two, | Template Table | | Table I.2-2 | Specific |
| three and all 4 antigens 3.1.2. Secondary objectives Table I – 3 CD4+ T cells expressing at least 2 | Template Table | | Table 12.2 | 0/ OMI |
| cytokines including IL-2 : Descriptive statistics Table I – 4 CD4+ T cells expressing at least 2 cytokines including IL-2 : Number and | I - 3 Template Table | | Table I.2-3 Table I.2-4 | %CMI<br>specific |
| percentage of responders per antigen Table I – 5 CD4+ T cells expressing at least 2 cytokines including IL-2: Number and percentage of responders to one, two, three or four antigens | Template Table<br>I - 5 | | Table I.2-5 | specific |
| Table I – 6 CD4+ T cells expressing at least 2 cytokines including IL-2: Number and percentage of responders to one, two, three or four antigens with specification of antigens | Template Table<br>I - 6 | | Supplementary<br>Table I.2-6 | specific |
| Table I – 7 CD4+ T cells expressing at least 2 cytokines including TNF- $\alpha$ : Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-7 | %CMI |
| Table I – 8 CD4+ T cells expressing at least 2 cytokines including IFN-γ: Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-8 | %CMI |
| Table I – 9 CD4+ T cells expressing at least 2 cytokines including CD40-L : Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-9 | %CMI |
| Table I – 10 CD4+ T cells expressing at least 2 cytokines : Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-10 | %CMI |
| 3.1.3. Exploratory objectives Table I – 1b Frequency of CD8+ T-cells | Template Table | | Working Table | Cuc-:E- |

1-1

Template Table

1-3

Template Table

1-3

expressing cytokines (by ICS) at pre-

statistics (amendment 1)

vaccination: percentiles (amendment 1) Table I - 11 CD8+ T cells expressing at least

α : Descriptive statistics (amendment 1)

one cytokine (TNF-α and/or IFN-γ): Descriptive

Table I - 12 CD8+ T cells expressing only TNF-

Specific

%CMI

%CMI

I.2-1b

Supplementary

Table I.2-11

Supplementary

Table I.2-12



| Denomination | Template table | Total<br>vaccinated<br>cohort | ATP cohort for immunogenicity | Macro |
|---|---|---|---|---|
| Table I – 13 CD8+ T cells expressing <b>only IFN-</b> γ: Descriptive statistics ( <b>amendment 1</b> ) | Template Table<br>I - 3 | | Supplementary<br>Table I.2-13 | %CMI |
| Table I – 14 CD8+ T cells expressing TNF-α and IFN-γ: Descriptive statistics (amendment 1) | Template Table<br>I - 3 | | Supplementary<br>Table I.2-14 | %CMI |
| Table I – 16 CD8+ T cells expressing at least one cytokine (TNF-α and/or IFN-γ): Number and percentage of responders per antigen (amendment 1) | Template Table<br>I - 4 | | Table I.2-16 | Specific |
| Table I – 17 CD4+ T cells expressing at least 2 cytokines including IL-2 (stimulaled with other HIV clade antigens): Descriptive statistics | Template Table<br>I - 3 | | Table I.2-17 | %CMI |
| Table I – 18 CD4+ T cells expressing at least 2 cytokines including TNF-α (stimulaled with other HIV clade antigens): Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-18 | %CMI |
| Table I – 19 CD4+ T cells expressing at least 2 cytokines including IFN-γ (stimulated with other HIV clade antigens): Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-19 | %CMI |
| Table I – 20 CD4+ T cells expressing at least 2 cytokines including CD40-L (stimulaled with other HIV clade Table I.2-4.antigens): Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-20 | %CMI |
| Table I – 21 CD4+ T cells expressing at least 2 cytokines (stimulaled with other HIV clade antigens): Descriptive statistics | Template Table<br>I - 3 | | Supplementary<br>Table I.2-21 | %CMI |
| 3.2. Antibodies by Elisa | | | | |
| Table I - 22 Seroposivity rates and GMTs for antibodies | Template Table<br>I - 7 | | Table I.2-22 | %GMT |

28

| gsk GlaxoSmithKline | Study RAP | |
|------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

# 5.3. Template of tables

# 5.3.1. Study cohorts and demography analysis

# 5.3.1.1. Study cohorts

Template Table D - 1 Number of subjects enrolled into the study as well as the number of subjects excluded from ATP analyses with reasons for exclusion

| | Total | Total | | | [Each group] |
|---------------------------|-------|-------|---|---|--------------|
| Title | n | S | % | n | s |
| Total enrolled cohort | | | | | |
| (code XXXX) | | | | | |
| Total vaccinated cohort | | | | | |
| (code XXXX) | | | | | |
| ATP safety cohort | | | | | |
| (code XXXX) | | | | | |
| ATP immunogenicity cohort | | | | | |

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the considered ATP cohort relative to the Total vaccinated cohort Data source = Appendix table IA

| gsk GlaxoSmithKline | | Study RAP | |
|---|---|---|---|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | ⊠ Final | Date: 26SEP 2008 |

# Template Table D - 2 Number of subjects at each visit and list of withdrawn subjects

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| [Each group] | VISIT 1 | | | |
| | VISIT 2 | | | |
| | VISIT 3 | | | |
| | VISIT 4 | | | |
| | VISIT 5 | | | |
| | VISIT 6 | | | |
| | VISIT 7 | | | |
| | VISIT 8 | | | |
| | VISIT 9 | | | |
| | VISIT 10 | | | |

Data source = Appendix table IC, Appendix table IEi

# Template Table D - 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal

| | [Each group] | Total |
|---|---|---|
| Number of subjects enrolled | | |
| Number of subjects completed | | |
| Number of subjects withdrawn | | |
| Reasons for withdraw: | | |
| Serious Adverse Event | | |
| Non-serious adverse event | | |
| Protocol violation | | |
| Consent withdrawal (not due to an adverse event) | | |
| Migrated/moved from study area | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | |
| Lost to follow-up (subjects with complete vaccination course) | | |
| Others | | |

Vaccinated = number of subjects who were vaccinated in the study Completed = number of subjects who completed last study visit Withdrawn = number of subjects who did not come for the last visit Data source = Appendix table IEi

#### Template Table D - 4 Minimum and maximum activity dates

| Activity number | | Minimum date | Maximum date |
|-----------------|--------------|--------------|--------------|
| [Each activity] | [Each visit] | DDMMMYYYY | DDMMMYYYY |
| | | DDMMMYYYY | DDMMMYYYY |

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

# Template Table D - 5 Number and pe

Number and percentage of subjects who received the vaccine dose(s)

| | [Each group]<br>(N =) | | tal<br>l =) |
|-----|-----------------------|---|-------------|
| | n % | n | % |
| 1 | | | |
| 2 | | | |
| Any | | | |

N = number of subjects in each group or in total included in the considered cohort

n/% = number/percentage of subjects receiving the specified total number of doses in each group or in total

Any = number and percentage of subjects receiving at least one dose

Data source = Appendix table IG, Appendix table IIA, Appendix table IIB

# Template Table D - 6 Deviations from specifications for age and intervals between study visits

| | | Age | VISIT 1 – VISIT 2 | [Other intervals] |
|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol |
| | | from xx to xx | From 0 to 0 days | from xx to xx days |
| [Each group] | N | | | |
| | n | | | |
| | % | | | |
| | range | | | |

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n/% = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

Data source = Appendix table IB, Appendix table ICi

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

#### 5.3.1.2. **Demographic characteristics**

#### Template Table D - 7 Summary of demographic characteristics

| | Parameters or | | roup] | Tot<br>N= | |
|---|---|---|---|---|---|
| Characteristics | Categories | Value or<br>n | % | Value<br>or n | % |
| Age(Years) | Mean<br>SD<br>Median<br>Minimum<br>Maximum | | | | |
| Gender | Female<br>Male | | | | |
| Race | African Heritage / African American American Indian or Alaskan Native Asian – Central / South Asian Heritage Asian – East Asian Heritage Asian – Japanese Heritage Asian – South East Asian Heritage Native Hawaiian or Other Pacific Islander White – Arabic / North African Heritage White – Caucasian / European Heritage Other | | | | |

N = number of subjects

n = number of subjects in a given category Value = value of the considered parameter

% = n/Number of subjects with available results x 100

Data source = Appendix table IB

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

# 5.3.2. Reactogenicity/Safety

# 5.3.2.1. Compliance with respect to documenting safety

#### Template Table R - 1 Compliance in returning symptom sheets

| Dose | | Number<br>Of | according | Of | Compliance<br>%<br>general | <br>Compliance<br>%<br>Local |
|---|---|---|---|---|---|---|
| 1 | [Each group] | | | | | |
| 2 | | | | | | |
| Total | | | | | | |

SS = Symptom sheets used for the collection of local and general solicited AEs
Compliance % = (number of doses with symptom sheet returned / number of administered doses) X 100
Data source = Appendix table IG, Appendix table IIA, Appendix table IIB

#### Template Table R - 2 Compliance to data capture

| | | [Each dose] | | [Each dose] All doses | | oses | Per subject |
|---|---|---|---|---|---|---|---|
| Group | Criteria | n | % | n | % | n | % |
| [Each group] | With visit done | | | | | | |
| | With dose received | | | | | | |
| | With local solicited data available | | | | | | |
| | With general solicited data available | | | | | | |
| Total | With visit done | | | | | | |
| | With dose received | | | | | | |
| | With local solicited data available | | | | | | |
| | With general solicited data available | | | | | | |

n = for each dose: number of subjects enrolled in the considered cohort and fulfilling specific criteria for the considered dose for all doses: sum of n from individual doses

per subject : number of subjects enrolled in the considered cohort and fulfilling specific criteria for at least one dose % = percentage of doses with solicited/unsolicited data available among the number of administered doses Data source = Appendix table IG

| gsk GlaxoSmithKline | Stu | dy RAP |
|--------------------------|--------------------|-------------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | n ⊠ Final | <b>Date:</b> 26SEP 2008 |

# 5.3.2.2. All symptoms

Template Table R - 3 Incidence and nature of symptoms reported during the 7-day (Days 0-6) post-vaccination period

| | | | Any Symptom | | General symptoms | | | | Local symptoms | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group | Ν | n | % | 95% | 6 CI | N | n | % | 95% | 6 CI | N | n | % | 95% | 6 CI |
| | | | | | LL | UL | | | | 님 | UL | | | | 님 | J |
| | [Each group] | | | | | | | | | | | | | | | |
| Dose 2 | [Each group] | | | | | | | | | | | | | | | |
| Overall/dose | [Each group] | | | | | | | | | | | | | | | |
| Overall/subj | [Each group] | | | | | | | | | | | | | | | |

For each dose and overall/subject:

N= number of subjects with at least one documented dose

n/%= number/percentage of subjects presenting at least one type of symptom whatever the study vaccine administered For overall/dose:

N= number of documented doses

n/%= number/percentage of doses followed by at least one type of symptom whatever the study vaccine administered 95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IIA, Appendix table IIB

| gsk GlaxoSmithKlir | ne | Study RAP | |
|---|---|---|---|
| Study Id: 10870 | 6 | Abbreviated Title: | PRO HIV-005 |
| Version: Dr | aft version | | <b>Date:</b> 26SEP 2008 |

# 5.3.2.3. Solicited symptoms

Template Table R - 4 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period

| | | | | [Each group] | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | 95 % | CI |
| Symptom | Follow-up | Туре | N | n | % | LL | UL |
| | | ch dose)/Overall dose/O | verall subject | | - | • | |
| Pain | <= 2 days | All | | | | | |
| | | Grade 3 | | | | | |
| | > 2 days | All | | | | | |
| Ī | | Grade 3 | | | | | |
| | Total | All | | | | | |
| | | Grade 3 | | | | | |
| Redness (mm) | <= 2 days | All | | | | | |
| | | > 20 | | | | | |
| | > 2 days | All | | | | | |
| | | > 20 | | | | | |
| | Total | All | | | | | |
| | | > 20 | | | | | $\top$ |
| Swelling (mm) | <= 2 days | All | | | | | |
| | | > 20 | | | | | |
| | > 2 days | All | | | | | |
| | • | > 20 | | | | | $\top$ |
| | Total | All | | | | | $\top$ |
| | | > 20 | | | | 1 | $\neg$ |

For each dose and overall/subject:

N= number of subjects with at least one documented dose

n/%= number/percentage of subjects reporting at least once the symptom For Overall/dose:

N= number of documented doses

n/%= number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Data source = Appendix table IIA

| gsk | SmithKline | Study RAP | |
|-----------|-----------------|--------------------|------------------|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | | Date: 26SEP 2008 |

Template Table R - 5

Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period

| | | | | [Each g | | | |
|---|---|---|---|---|---|---|---|
| | | | | - | | 95 % | CI |
| Symptom | Follow-up | Туре | N | n | % | LL | UL |
| | | | [E | ach dose | /Overall<br>subject | | Overall |
| (Each symptom) | <= 2 days | All | | | | | |
| | | Grade 3 | | | | | |
| | | Rel | | | | | |
| | | Rel*Grade 3 | | | | | |
| | > 2 days | All | | | | | |
| | | Grade 3 | | | | | |
| | | Rel | | | | | |
| | | Rel*Grade 3 | | | | | |
| | Total | All | | | | | |
| | | Grade 3 | | | | | |
| | | Rel | | | | | |
| | | Rel*Grade 3 | | | | | |

For each dose and overall/subject:

N= number of subjects with at least one documented dose

n/%= number/percentage of subjects reporting at least once the symptom

For Overall/dose:

N= number of documented doses

n/%= number/percentage of doses followed by at least one type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Data source = Appendix table IIB

# Template Table R - 6 Number of days with symptoms during the solicited post-vaccination period

| Solicited symptom | Dose | Group | N | Mean | Min | Q1 | Median | Q3 | Max |
|---|---|---|---|---|---|---|---|---|---|
| (Each symptom) | (Each dose) | [Each Group] | | | | | | | |
| | [Overall/dose] | | | | | | | | |

N = number of doses with the symptom

Q1 = 25th percentile

Q3 = 75th percentile

Data source = Appendix table IIA, Appendix table IIB

| gsk GlaxoSmithKline | Stu | dy RAP |
|------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

Template Table R - 7 Maximum temperature per dose, overall doses, overall subject (0.5° increments)

| | | | [] | Each gro | oup] | |
|---------|-----------------------|--------|------------|----------|------|----|
| | | 95 % ( | | | CI | |
| Symptom | Туре | N | n | % | LL | UL |
| | (Each dose)/Overall d | ose/Ov | erall subj | ect | | |
| Fever | All | | | | | |
| | 37.5 - 38.0°C | | | | | |
| | 38.1 - 38.5°C | | | | | |
| | 38.6 - 39.0°C | | | | | |
| | 39.1 - 39.5°C | | | | | |
| | 39.6 - 40.0°C | | | | | |
| | 40.1°C + | | | | | |
| | Rel*[37.5 - 38.0°C[ | | | | | |
| | Rel* [38.1 - 38.5°C[ | | | | | |
| | Rel* [38.6 - 39.0°C[ | | | | | |
| | Rel* [39.1 - 39.5°C[ | | | | | |
| | Rel* [39.6 - 40.0°C[ | | | | | |
| | Rel* [40.1°C[ | | | | | |

For each dose and overall/subject:

N= number of subjects with at least one documented dose

n/%= number/percentage of subjects reporting at least once the symptom

For Overall/dose:

N= number of documented doses

n/%= number/percentage of doses followed by at least one type of symptom 95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Data source = Appendix table IIB

| <b>gsk</b> GlaxoSmithKline | St | tudy RAP |
|----------------------------|--------------------|------------------|
| Study Id: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft versi | on ⊠ Final | Date: 26SEP 2008 |

# 5.3.2.4. Unsolicited symptoms

Template Table R - 8

Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 0-29) post-vaccination period

| System | Preferred | [Each group] (N=) | | | |
|---|---|---|---|---|---|
| Organ Class | Term | n | % | 95%CI | |
| (CODE) | (CODE) | | | LL | UL |
| At least one symptom | | | | | |
| [Each SOC] | [Each preferred term] | | | | |

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of administered doses

n/% = number/percentage of doses with the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IICi

| <b>gsk</b> GlaxoSmithKline | Stu | dy RAP |
|----------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

Template Table R - 9

Percentage of doses with unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, within the 30-day (Days 0-29) post-vaccination period

| System | Preferred | [Each group] (N=) | | | |
|---|---|---|---|---|---|
| Organ Class | Term | n | % | 95%CI | |
| (CODE) | (CODE) | | | LL | UL |
| At least one symptom | | | | | |
| [Each SOC] | [Each preferred term] | | | | |

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of administered doses

n/% = number/percentage of doses with the symptom

95% CI= exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IICi

# Template Table R - 10 Global Summary of unsolicited signs and symptoms reported within the 30-day (Days 0-29) post-vaccination period

| | [Each group] | Total |
|---|---|---|
| Number of subjects with at least one unsolicited symptom reported | | |
| Number of doses followed by at least one unsolicited symptom | | |
| Number of unsolicited symptoms classified by MEDDRA Preferred | | |
| Term* | | |
| Number of unsolicited symptoms reported | | |

<sup>\*</sup> Symptoms reported by a subject after a given dose and classified by the same Preferred Term are counted once Data source = Appendix table IICi

38

| gsk GlaxoSmithKline | Stu | dy RAP |
|--------------------------|--------------------|------------------|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | ☑ Final | Date: 26SEP 2008 |

#### 5.3.2.5. Serious adverse events

Template Table R - 11 Listing of SAEs

| | • | Sub.<br>No. | Case<br>Id | Age<br>at<br>onset<br>(Year) | Verbatim | Preferred<br>term | System<br>Organ<br>Class | MA<br>type | Dose | Day<br>of<br>onset | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ŀ | | | | (Toul) | | | | | | OHIOCE | | |
| Į | | | | | | | | | | | | |

<sup>\* =</sup> SAEs available in OCEAN but not in Clinical Data Base

## 5.3.2.6. Haematology and biochemistry

# Template Table R - 12 Distribution of haematology and biochemistry with respect to normal laboratory ranges

| | [Each group] | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | -UnkBelow- | | -Within- | | -Above- | | | |
| Laboratory parameter | Timing | N | n | % | n | % | n | % | n | % |
| [Each parameter] | [Each timing] | | | | | | | | | |

Unk. = Laboratory value unknown

% = Percentage of subjects based on N

N = total number of subjects with available results

n = Number of subjects in the appropriate category

Data source = Appendix table IV.a, IV.B

# Template Table R - 13 Change from baseline in hematological and biochemical levels with respect to normal ranges

| | | | [Each group] | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | -Be | low- | -Wit | thin- | -Ab | ove- | -Alert- | |
| Laboratory | Timing | Baseline | N | n | % | n | % | n | % | n | % |
| parameter | | Assessment | | | | | | | | | |
| [Each laboratory parameter] | [Each timing] | Below | | | | | | | | | |
| | | Within | | | | | | | | | |
| | | Above | | | | | | | | | |
| | | Alert | | | | | | | | | |

N = number of subjects with available results

n/% = number/percentage of subjects in the specified category

Data source = Appendix table IV.a, IV.B

<sup>???????? =</sup> SAEs available in Clinical Data Base but not in OCEAN

| <b>gsk</b> GlaxoSmithKline | Study RAP | |
|---|---|---|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |

#### 5.3.2.7. Concomitant medications

Template Table R - 14 Incidence of concomitant medication during the 30-day (Days 0-29) post-vaccination period

| | | [Eac | h group | 0] | |
|---|---|---|---|---|---|
| | | | | 95% | 6 CI |
| | N | n | % | LL | UL |
| [Each dose] [Overall/dose] [Overall/subject] | | | | | |
| Any | | | | | |
| Any antibiotic | | | | | |
| Any antipyretic | | | | | |
| Any immunosuppressant | | · | | | |

For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects who started to take the specified concomitant medication at least once during the mentioned period

For overall/dose:

N= number of administered doses

n/%= number/percentage of doses after which the specified concomitant medication was started at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IIDi

| gsk GlaxoSmithKline | Study RAP | |
|---|---|---|
| Study ld: 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: Draft version | on 🗵 Final | Date: 26SEP 2008 |

## 5.3.3. Immunogenicity

#### 5.3.3.1. CD4+/CD8+ T-cells response by ICS

Template Table I - 1 Frequency of CD4+/CD8+ T-cells expressing cytokines (by ICS) at pre-vaccination: Percentiles

| Type of | Antigen | Cytokines | Percentiles | | | |
|---|---|---|---|---|---|---|
| T-cells | | | 90% | 95% | 99% | 100% |
| [CD4+ or<br>CD8+] | [ p17 or p24<br>or Nef or Tat<br>or F4Co ] | | | | | |

Data source = Appendix table IIIB

# Template Table I - 2

Frequency of CD4+/CD8+ T-cells expressing cytokines (ICS): Number and percentage of responders to at least one, two, three and all 4 antigens

| Group | Timing | Number of<br>antigens | N | n | % | 95% | 6 CI |
|---|---|---|---|---|---|---|---|
| | | unagono | | | | LL | UL |
| [Each group] | [Each Timing] | At least 1 antigen | | | | | |
| | | At least 2 antigens | | | | | |
| | | At least 3 antigens | | | | | |
| | | All 4 antigens | | | | | |

N = number of subjects with available results for all 4 antigens (amendment 1)

n/% = number/percentage of subjects in the specified category

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IIIB

# Template Table I - 3

Frequency of CD4+/CD8+ T-cells expressing cytokines (ICS) : Descriptive statistics

| Stimulating Ag | Study Group | Activity | N | Mean | SD | Min | Q1 | Median | Q3 | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| [Each stimulation] | [Each group] | [Each timing] | | | | | | | | |

N = number of subjects with available results

SD= standard deviation

Q1/Q3 = first/third quartile

MIN/MAX = Minimum/Maximum

Data source = Appendix IIIB

| gsk | SmithKline | Study RAP | |
|---|---|---|---|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | ⊠ Final | Date: 26SEP 2008 |

Template Table I - 4

Frequency of CD4+/CD8+ T-cells expressing cytokines (ICS) : Number and percentage of responders per antigen

| Group | Timing | Antigens | N | n | % | 95% CI | |
|--------------|---------------|----------|---|---|---|--------|----|
| | | | | | | LL | UL |
| [Each group] | [Each Timing] | p17 | | | | | |
| | | p24 | | | | | |
| | | Nef | | | | | |
| | | RT | | | | | |

N = number of subjects with available results n/% = number/percentage of subjects in the specified category

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IIIB

#### Template Table I - 5

Frequency of CD4+/CD8+ T-cells expressing cytokines (ICS): Number and percentage of responders to one, two, three or four antigens

| Group | Timing | Number of<br>antigens | N | n | % | 95% | % CI |
|---|---|---|---|---|---|---|---|
| | | anagens | | | | LL | UL |
| [Each group] | [Each Timing] | None | | | | | |
| | | 1 antigen | | | | | |
| | | 2 antigens | | | | | |
| | | 3 antigens | | | | | |
| | | 4 antigens | | | | | |

N = number of subjects with available results for all 4 antigens (amendment 1)

n/% = number/percentage of subjects in the specified category

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IIIB

| gsk | SmithKline | Study RAP | |
|---|---|---|---|
| Study Id: | 108706 | Abbreviated Title: | PRO HIV-005 |
| Version: | ☐ Draft version | ⊠ Final | Date: 26SEP 2008 |

Template Table I - 6

Frequency of CD4+/CD8+ T-cells expressing cytokines (ICS): Number and percentage of responders to one, two, three or four antigens with specification of antigens

| | Timing | Number of antigens | | | n | % | 95% CI | |
|---|---|---|---|---|---|---|---|---|
| Group | | | Ag Stimulation | N | | | LL | UL |
| [Each group] | [Each timing] | None | None | | | | | |
| | | | Any | | | | | |
| | | 1 antigen | p17 | | | | | |
| | | | [other] | | | | | |
| | | 2 antigens Any p17+p24 [other] | Any | | | | | |
| | | | p17+p24 | | | | | |
| | | | [other] | | | | | |
| | | | Any | | | | | |
| | | 3 antigens | p17+p24+Nef | | | | | |
| | | | [other] | | | | | |
| | | 4 antigens | p17+p24+Nef+RT | | | | | |

N = number of subjects with available results for all 4 antigens (amendment 1)

n/% = number/percentage of subjects with a number of expressed cells above or equal the cut-off

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Data source = Appendix table IIIB

#### 5.3.3.2. Antibodies

#### Template Table I - 7 Seropositivity rates and GMT for each antibody

| | | | | | >=cut-off | | | GMT | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | % CI | | 95% | 6 CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| [Each antibody] | [Each group] | [Each timing] | | | | | | | | | | |

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with concentration within the specified range

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

MIN/MAX = Minimum/Maximum

Data source = Appendix table IIIA